CLINICAL TRIAL: NCT06313502
Title: High Dose Ascorbic Acid (HDAA) in Patients With Plasma Cell Disorders
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 274271
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Plasma Cell Disorder
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 75gm HDAA + Melphalan 100mg/m2 (Experimental): Subjects will receive HDAA alone (75gm) on day -4, HDAA combined with melphalan 100 mg/m2 on day -1, and ASCT on day 0. Four additional HDAA doses (75gm) will then be administered 3 days apart on D+2, D+5, D+8 and D+11, followed by weekly doses of the corresponding dose of HDAA for four additional weeks. On day, D-1, when both drugs are given, melphalan should be given first
  Interventions: Drug: 75gm HDAA
- 100gm HDAA + Melphalan 100mg/m2 (Experimental): Subjects will receive HDAA alone (100gm) on day -4, HDAA combined with melphalan 100 mg/m2 on day -1, and ASCT on day 0. Four additional HDAA doses (100gm) will then be administered 3 days apart on D+2, D+5, D+8 and D+11, followed by weekly doses of the corresponding dose of HDAA for four additional weeks. On day, D-1, when both drugs are given, melphalan should be given first
  Interventions: Drug: 100gm HDAA
- 125gm HDAA + Melphalan 100mg/m2 (Experimental): Subjects will receive HDAA alone (125gm) on day -4, HDAA combined with melphalan 100 mg/m2 on day -1, and ASCT on day 0. Four additional HDAA doses (125gm) will then be administered 3 days apart on D+2, D+5, D+8 and D+11, followed by weekly doses of the corresponding dose of HDAA for four additional weeks. On day, D-1, when both drugs are given, melphalan should be given first
  Interventions: Drug: 125gm HDAA

INTERVENTIONS:
Drug: 75gm HDAA — Initiation: Subjects will receive a test dose of ascorbate (15 gm), during screening period, prior to starting therapy.
  Dose: After successfully completing the test dose, subjects will receive 75gm of ascorbate infusion. Dose modifications will not be made for weight or body surface area.
  Administration: Infusion time is set to occur at 120 minutes +/-10 minutes but may be adjusted for subject comfort. The infusion rate should not exceed 500 mL/hour without consulting with PI. Changes in infusion rates should be recorded.
  Arms: 75gm HDAA + Melphalan 100mg/m2
Drug: 100gm HDAA — Initiation: Subjects will receive a test dose of ascorbate (15 gm), during screening period, prior to starting therapy.
  Dose: After successfully completing the test dose, subjects will receive 100gm of ascorbate infusion. Dose modifications will not be made for weight or body surface area.
  Administration: Infusion time is set to occur at 180 minutes +/-10 minutes but may be adjusted for subject comfort. The infusion rate should not exceed 500 mL/hour without consulting with PI. Changes in infusion rates should be recorded.
  Arms: 100gm HDAA + Melphalan 100mg/m2
Drug: 125gm HDAA — Initiation: Subjects will receive a test dose of ascorbate (15 gm), during screening period, prior to starting therapy.
  Dose: After successfully completing the test dose, subjects will receive 125gm of ascorbate infusion. Dose modifications will not be made for weight or body surface area.
  Administration: Infusion time is set to occur at 240 minutes +/-10 minutes but may be adjusted for subject comfort. The infusion rate should not exceed 500 mL/hour without consulting with PI. Changes in infusion rates should be recorded.
  Arms: 125gm HDAA + Melphalan 100mg/m2

SUMMARY:
The purpose of this research is to evaluate whether HDAA in combination with a single dose of 100 mg/m2 IV melphalan followed by autologous stem cell transplantation (ASCT) is safe and effective for subjects with relapsed refractory multiple myeloma. The proposed melphalan dose is 50% of the current standard myeloablative dose (200 mg/m2). Based on our preclinical data, the investigator hypothesize that the combination of reduced dose melphalan with IV HDAA will have high efficacy and tolerability

Primary Objective To determine tumor response using International Myeloma Working Group (IMWG) criteria (see Appendix B).

Secondary Objectives

Objectives:

1. Determine the safety and tolerability of HDAA in combination with reduced dose melphalan conditioning and autologous stem cell transplantation (ASCT) in relapsed refractory multiple myeloma subjects.
2. Determine the rate of Minimal Residual Disease (MRD) negativity at time point of response assessment using 8 color flow cytometry on BM sample. Functional imaging, such as positron emission tomography (PET) scan and magnetic resonance imaging (MRI), will also be performed to assess the disease status.
3. Categorize and quantify adverse events compared to historical control.
4. Determine quality of life parameters using standardized health-related quality of life measures
5. Determine oxidative stress parameters in plasma during treatment.

DETAILED DESCRIPTION:
This is a single arm Phase I trial evaluating safety, tolerability, and efficacy of High Dose Ascorbic Acid (HDAA) in patients with plasma cell disorders. This is a single arm study. Subjects will receive a test dose of HDAA alone at screening (15gm), then proceed to either 75, 100, or 125 gm, depending upon the cohort) on day -4, HDAA combined with melphalan 100 mg/m2 on day -1, and ASCT on day 0. Four additional HDAA doses (each of which is either 75, 100, or 125 gm, depending upon the cohort) will then be administered 3 days apart on D+2, D+5, D+8 and D+11, followed by weekly doses of the corresponding dose of HDAA for four additional weeks.Lab tests, vitals, and scans will be performed to assess tolerability, safety, and efficacy at each scheduled infusion timepoint.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent.
2. Participants who are 18 years of age or older
3. Subjects who have been previously treated with 3 or more lines of therapy (i.e., proteasome inhibitors, immunomodulatory agents such as lenalidomide, and monoclonal antibodies such as daratumumab) and have progressed within past 6 months.
4. Subjects who have at least 1x106/kg CD34 stem cells in storage
5. Subjects must have measurable disease (as determined by the UAMS clinical lab), including at least one of the criteria below. Tests performed as SOC within 30 days of the first dose may be utilized:

   * M-protein quantities ≥ 0.5 gm/dl by SPEP
   * ≥ 200 mg/24-hour urine collection by UPEP
   * serum-free light chain levels > 100 mg/L (milligrams/liter involved light chain) and an abnormal kappa/lambda (κ/λ) ratio in subjects without detectable serum or urine m-protein
   * a serum IgA level ≥ 500 mg/dL for subjects with immunoglobulin class A (IgA) myeloma whose disease can only be reliably measured by quantitative immunoglobulin measurement
   * Non-secretory subjects are eligible provided the subject has > 20% BM plasmacytosis, OR multiple plasmacytomas or lesions (≥3) on MRI at the time of diagnosis or study enrollment, OR the presence of lesions (≥ 3) on PET/Computerized Tomography (CT) scan.
6. Adequate organ function reflects the following:

   * Absolute neutrophil count (ANC) ≥ 0.5 x 109/L without growth factor support for 7 days (14 days if pegfilgastrim).
   * Platelets ≥ 25 x 109/L without transfusion for 7 days. However, subject can be enrolled if the ANC and platelets are low due to disease
   * Potassium within normal limits or correctable with supplements
   * Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x upper limit of normal (ULN)
   * Serum bilirubin ≤ 1.5 x ULN
   * Estimated serum creatinine clearance of ≥ 45 mL/min using the Cockcroft-Gault equation or directly calculated from the 24-hour urine collection method
   * International normalized ratio (INR) < 1.5 x ULN and partial thromboplastin time < 1.5 x ULN
   * Ejection fraction by ECHO or MUGA of ≥ 40% performed
   * Subjects must have adequate pulmonary function studies (PFTs) > 50% of predicted on mechanical aspects (forced expiratory volume, forced vital capacity) and > 50% of predicted (adjusted for hemoglobin) on diffusion capacity. If the participant is unable to complete PFTs due to disease-related pain or other circumstances that make it difficult to reliably perform PFTs, documentation of pulmonary function adequate for transplant will occur via a CT scan without evidence of major pulmonary disease and arterial blood gas results.
7. Subjects must have a performance status of 0-2 based on ECOG performance criteria. Subjects with poor performance status (3-4) based solely on bone pain will be eligible if there is documentation to verify this.
8. Negative serum or urine pregnancy test (sensitivity of at least 25 mIU/mL) at screening.

Exclusion Criteria:

1. Prior allogeneic transplant.
2. Known hypersensitivity or allergy to ascorbic acid or melphalan, or any Grade 3 or higher AE as a result of test dose given during screening (15 gm).
3. Subjects must not have a concurrent malignancy unless it can be adequately treated by non-chemotherapeutic intervention. Participants may have a history of prior malignancy without any chemotherapy within 365 days of study entry AND life expectancy exceeding 5 years at the time of study entry.
4. Subjects must not have life-threatening comorbidities as assessed by the investigator.
5. History or evidence of MM associated with immunodeficiency states (e.g., hereditary immune deficiency, human immunodeficiency virus (HIV), organ transplant, or leukemia).
6. Known HIV disease (requires negative test for clinically suspected HIV infection).
7. Evidence of CNS myeloma.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, recent (within 6 months) myocardial infarction, uncontrolled or symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension on appropriate therapy or psychiatric illness/social situations that would limit compliance with study requirements.
9. Concurrent use of coumadin (warfarin).
10. Glucose-6-phosphate dehydrogenase deficiency as defined by blood test at screening visit.
11. Pre-existing renal insufficiency or renal failure, a known history of renal stones, or who are undergoing dialysis.
12. Diabetic subjects who are insulin dependent.
13. Any other condition that, in the opinion of the investigator, might interfere with the safe conduct of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Tumor Response measured by IMWG criteria | End of Treatment (approx. 24 months from beginning of enrollment)
  To determine tumor response using International Myeloma Working Group (IMWG) criteria

SECONDARY OUTCOMES:
Safety and Tolerability of HDAA with reduced dose melphalan measured using number and severity of AEs | End of Treatment (approx. 24 months from beginning of enrollment)
  The number and severity of all AEs will be summarized by simple descriptive statistics and compared to a historical control.
Rate of Minimal Residual Disease (MRD) negativity using 8 color flow cytometry | End of Treatment (approx. 24 months from beginning of enrollment)
  8 color flow cytometry on BM sample, functional imaging, such as positron emission tomography (PET) scan and magnetic resonance imaging (MRI), will also be performed to assess the disease status.
Determine quality of life parameter using QLQ-C30 | End of Treatment (approx. 24 months from beginning of enrollment)
  Determined using standardized health-related quality of life measures.
Determine quality of life parameter using EQ-5D-5L | End of Treatment (approx. 24 months from beginning of enrollment)
  Determined using standardized health-related quality of life measures.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Schinke, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States